CLINICAL TRIAL: NCT03311126
Title: Bendamustine + Obinutuzumab Induction Chemoimmunotherapy With Risk-adapted Obinutuzumab Maintenance Therapy in Previously Untreated Mantle Cell Lymphoma
Brief Title: Bendamustine + Obinutuzumab Induction With Obinutuzumab Maintenance in Untreated Mantle Cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW16086; 2017-0609 (Other: Institutional Review Board); NCI-2017-01729 (Registry Identifier: NCI CTRP); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison); Protocol Version 11/18/2019 (Other: UW Madison)
Record Dates: First submitted 2017-09-28; First posted 2017-10-16 (Actual); Results first posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Mantle Cell Lymphoma; Non-hodgkin Lymphoma; Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma, Non-Hodgkin | interventions — Bendamustine Hydrochloride; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bendamustine + Obinutuzumab (BO) (Experimental): Induction chemoimmunotherapy (28 day cycles):
  Bendamustine 90 mg/m2 IV days 1 & 2 every 28 days X 4-6 cycles
  Obinutuzumab:
  * Cycle 1: 100 mg IV day 1, 900 mg IV day 2, 1000 mg IV days 8 & 15
  * Cycles 2-6: 1000 mg IV day 1
  Consolidation phase:
  Obinutuzumab 1000 mg IV weekly X 4 doses
  Maintenance phase (8 week cycles):
  Obinutuzumab 1000 mg IV on day 1 of cycles 1-8
  Interventions: Drug: Bendamustine; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Bendamustine — Bendamustine is a chemotherapeutic agent that has dual functional properties of both an alkylating agent and a nitrogen mustard. Through these unique cytostatic properties, bendamustine is able to inhibit DNA transcription, replication, and repair. Bendamustine is approved in the U.S. for treatment of chronic lymphocytic leukemia (CLL) and for indolent B cell non-Hodgkin lymphomas (NHLs) progressing during or within 6 months of rituximab or a rituximab - containing regimen.
Drug: Obinutuzumab — Obinutuzumab is a glycoengineered, humanized, type II anti-CD20 monoclonal antibody (mAb).
  Other Names: GA101; RO5072759

SUMMARY:
This is a phase II single-arm, open-label, multicenter study evaluating the efficacy and safety of the combination of induction chemoimmunotherapy with bendamustine and obinutuzumab (BO) followed by consolidation therapy and maintenance therapy with obinutuzumab in subjects who have not received prior cytotoxic chemotherapy for their Mantle Cell Lymphoma (MCL) (i.e., prior single agent rituximab is permitted, prior involved-field radiotherapy is permitted).

DETAILED DESCRIPTION:
This is a phase II single-arm, open-label, multicenter study evaluating the efficacy and safety of the combination of induction chemoimmunotherapy with bendamustine and obinutuzumab (BO) followed by consolidation therapy and maintenance therapy with obinutuzumab in subjects who have not received prior cytotoxic chemotherapy for their MCL (i.e., prior single-agent rituximab is permitted, prior involved-field radiotherapy is permitted). Therapy for individual subjects will be risk-adapted based on results of minimal residual disease (MRD) testing performed after the consolidation phase. The study will be carried out at the University of Wisconsin Carbone Cancer Center (UWCCC) and participating community and academic practice sites within the Wisconsin Oncology Network (WON). There will be 6-10 sites participating in this study.

The subject participation will include a screening period, treatment period, and a follow-up period. The induction chemoimmunotherapy regimen consists of bendamustine and obinutuzumab for 4-6 cycles, followed by consolidation and maintenance therapy with obinutuzumab in subjects achieving an objective response to induction therapy (i.e., complete or partial response; stable disease with objective evidence of tumor shrinkage. Subjects who are MRD-negative (determined by MRD testing on bone marrow and PB) after consolidation therapy will omit maintenance therapy.

Subjects will undergo disease reassessment after C4 of induction BO chemoimmunotherapy, after obinutuzumab consolidation therapy, and after C4 and C8 of maintenance obinutuzumab. MRD testing will be done after C2 of induction (PB only), after consolidation (BMA and PB), and post-maintenance or end of treatment (EOT) (PB only).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the time of signing the informed consent document.
2. Histologically confirmed mantle cell lymphoma (confirmation of cyclin D1 positivity on diagnostic biopsy).
3. Subjects must have at least one bi-dimensionally measurable lesion; one of the measurements must be ≥1.5 cm in one direction
4. No prior cytotoxic chemotherapy; prior therapy with single-agent rituximab is permitted. Prior involved-field radiotherapy to symptomatic nodal sites of involvement is also permitted.
5. Prior therapy with rituximab is permitted, even in the setting of rituximab-refractory disease.
6. Must meet one of the following criteria:

   1. Not eligible for more intensive cytotoxic chemotherapy or consolidative autologous stem cell transplant based on one or more of the following:

      * Clinically significant heart or lung comorbidities, as reflected by at least 1 of the following:

        * Left ventricular ejection fraction (LVEF) ≤ 50%
        * Chronic stable angina or congestive heart failure controlled with medication
        * New York Heart Association (NYHA) class III or IV heart failure
        * Symptomatic chronic pulmonary disease or requirement for intermittent or continuous oxygen therapy
      * Presence of other medical comorbidity or limitation in functional status which the investigator judges to be incompatible with an acceptable risk to the subject with the use of intensive chemotherapy. The associated comorbidity or functional limitation must be clearly documented in the medical record at the time of enrollment.

      OR
   2. Subject has been informed of the risks and benefits of intensive chemotherapy and autologous stem cell transplant for treatment of mantle cell lymphoma and has refused this option. This discussion must be clearly documented in the medical record at the time of enrollment.
7. Eastern Cooperative Oncology Group (ECOG) performance status of ≤2 at study entry.
8. Laboratory test results within these ranges:

   1. Absolute neutrophil count ≥1500/µL.
   2. Platelet count ≥100,000/µL.
   3. Subjects with neutrophils <1500/µL or platelets <100,000/µL with splenomegaly or extensive bone marrow involvement as the etiology for their cytopenias are eligible.
   4. Subjects must have adequate renal function with a creatinine clearance of ≥40 mL/min as determined by the Cockcroft-Gault calculation.
   5. Total bilirubin ≤2X upper limit laboratory normal (ULN); subjects with nonclinically significant elevations of bilirubin due to Gilbert's disease are not required to meet these criteria.
   6. Serum transaminases AST (SGOT) and ALT (SGPT) ≤5X ULN.
   7. Serum alkaline phosphatase ≤5X ULN.
9. Disease-free of prior malignancies for ≥2 years with the exception of basal or squamous cell skin carcinoma, carcinoma "in situ" of the breast or cervix, or localized prostate cancer (treated definitively with hormone therapy, radiotherapy, or surgery).
10. Life expectancy of at least 3 months.
11. Understand and voluntarily sign an informed consent document.

Exclusion Criteria:

1. Subjects are not eligible if there is a prior history or current evidence of central nervous system or leptomeningeal involvement.
2. Concurrent use of other anti-cancer agents or treatments.
3. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent document or complying with the protocol treatment.
4. Prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical or breast cancer, or other cancer from which the subject has been disease free for at least 2 years.
5. Severe or life-threatening anaphylaxis or hypersensitivity reaction when previously exposed to rituximab or other mAb therapy.
6. Known to be positive for HIV or infectious hepatitis (type B or C).
7. Pregnant or breast-feeding females.
8. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Chang, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UW Carbone Cancer Center home page — http://www.uwhealth.org/uw-carbone-cancer-center/47424

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at UW Hospital and Clinics in Madison, WI, UW Cancer Center at ProHealth in Waukesha, WI, and St. Vincent Regional Cancer Center in Green Bay, WI from September 2017 to January 2022.
Groups:
- Bendamustine + Obinutuzumab (BO): Induction chemoimmunotherapy (28 day cycles):
  Bendamustine 90 mg/m2 IV days 1 & 2 every 28 days X 4-6 cycles
  Obinutuzumab:
  * Cycle 1: 100 mg IV day 1, 900 mg IV day 2, 1000 mg IV days 8 & 15
  * Cycles 2-6: 1000 mg IV day 1
  Consolidation phase:
  Obinutuzumab 1000 mg IV weekly X 4 doses
  Maintenance phase (8 week cycles):
  Obinutuzumab 1000 mg IV on day 1 of cycles 1-8
  Bendamustine: Bendamustine is a chemotherapeutic agent that has dual functional properties of both an alkylating agent and a nitrogen mustard. Through these unique cytostatic properties, bendamustine is able to inhibit DNA transcription, replication, and repair. Bendamustine is approved in the U.S. for treatment of chronic lymphocytic leukemia (CLL) and for indolent B cell non-Hodgkin lymphomas (NHLs) progressing during or within 6 months of rituximab or a rituximab - containing regimen.
  Obinutuzumab: Obinutuzumab is a glycoengineered, humanized, type II anti-CD20 monoclonal antibodies (mAb).
Period: Induction
Arm/Group | Bendamustine + Obinutuzumab (BO)
Started | 21
Induction Chemotherapy Cycle 4 | 21
Completed | 20
Not Completed | 1
Not completed — Death | 1
Period: Consolidation
Arm/Group | Bendamustine + Obinutuzumab (BO)
Started | 20
Completed | 20
Not Completed | 0
Period: Restaging Imaging
Arm/Group | Bendamustine + Obinutuzumab (BO)
Started | 20
Radiographic Complete Response | 10
Lack of Radiographic Complete Response | 10
Completed | 10
Not Completed | 10
Not completed — Radiographic Complete Response moved to Observation rather than Maintenance | 10
Period: Maintenance
Arm/Group | Bendamustine + Obinutuzumab (BO)
Started | 10
Discontinued Maintenance Early | 6
Completed All 8 Cycles | 4
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Bendamustine + Obinutuzumab (BO): Induction chemoimmunotherapy (28 day cycles):
  Bendamustine 90 mg/m2 IV days 1 & 2 every 28 days X 4-6 cycles
  Obinutuzumab:
  * Cycle 1: 100 mg IV day 1, 900 mg IV day 2, 1000 mg IV days 8 & 15
  * Cycles 2-6: 1000 mg IV day 1
  Consolidation phase:
  Obinutuzumab 1000 mg IV weekly X 4 doses
  Maintenance phase (8 week cycles):
  Obinutuzumab 1000 mg IV on day 1 of cycles 1-8
  Bendamustine: Bendamustine is a chemotherapeutic agent that has dual functional properties of both an alkylating agent and a nitrogen mustard. Through these unique cytostatic properties, bendamustine is able to inhibit DNA transcription, replication, and repair. Bendamustine is approved in the U.S. for treatment of CLL and for indolent B cell NHLs progressing during or within 6 months of rituximab or a rituximab - containing regimen.
  Obinutuzumab: Obinutuzumab is a glycoengineered, humanized, type II anti-CD20 mAb.
Arm/Group | Bendamustine + Obinutuzumab (BO)
Number analyzed (Participants) | 21
Age, Customized [Count of Participants; unit: Participants]
  50-59 years | 1
  60-69 years | 8
  70-79 years | 9
  80-89 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 means fully active, no restrictions, 1 means restricted in physically strenuous activity and able to carry out light activity, 2 means able to walk and capable of self-care but not work activities - up and about more than half of waking hours.
  Participants
    ECOG Performance Status 0 | 9
    ECOG Performance Status 1 | 9
    ECOG Performance Status 2 | 3
Stage [Count of Participants; unit: Participants] — Stage II cancer is large and contained in the organ it started in, Stage III cancer has grown into nearby tissues, and Stage IV cancer has spread to other parts of the body.
  Participants
    Stage II | 1
    Stage III | 0
    Stage IV | 20
MIPI Score [Count of Participants; unit: Participants] — Mantle Cell Lymphoma International Prognostic Index (MIPI) combines age, performance status, lactate dehydrogenase (LDH), and leukocyte count to identify low, intermediate, and high risk groups.
  Participants
    Low Risk | 1
    Intermediate Risk | 6
    High Risk | 14
Prior Treatment [Count of Participants; unit: Participants] — prior involved-site radiotherapy
  Participants | 1
Bulky Nodes [Count of Participants; unit: Participants] — Greater than 5 centimeters
  Participants | 7
Marrow Involvement [Count of Participants; unit: Participants] | 20
LDH elevation [Count of Participants; unit: Participants] | 9
Splenomegaly [Count of Participants; unit: Participants] — Enlargement of the spleen
  Participants | 10
P53 mutation status [Count of Participants; unit: Participants] — Population: number of participants with confirmed p53 testing
  Participants
    number analyzed (Participants) | 12
    (all) | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) at 2 Years
Description: For each patient, progression-free survival (PFS) is measured from cycle 1 day 1 (C1D1) of induction chemoimmunotherapy to the day patient experiences an event of disease progression or death, whichever occurs first. If a patient has not experienced an event at the time of analysis, patient's data will be censored at the date of the last available evaluation. The 2-year PFS probability will be estimated using the Kaplan-Meier method. From the date of C1D1 of induction therapy to the date of progression or death; in the absence of progression or death, participants will be followed for a minimum of 24 months after completion of study-related treatment. PFS rates at 2 years are reported here.
Time Frame: Up to 2 years
Measure: Number (95% Confidence Interval); unit: percent participants
Arm/Group | Bendamustine + Obinutuzumab (BO)
Number analyzed (Participants) | 21
percent participants | 66 [41.6 to 82.2]

2. Secondary Outcome: Minimal Residual Disease (MRD) Status
Description: MRD defined as reduction to >=10^-6 fold reduction in the IgVH unique clone of mantle cell lymphoma (MCL) by next generation (NGS).
  MRD status will be evaluated after 2 cycles of induction chemoimmunotherapy with bendamustine and obinutuzumab, after 4 cycles of consolidation with obinutuzumab, and after an additional 8 cycles of maintenance with obinutuzumab. MRD status will be summarized using frequency and proportion with 95% confidence intervals.
  MRD status will be collected on peripheral blood after cycle 2 of induction therapy, on peripheral blood and bone marrow aspirate after consolidation obinutuzumab, and peripheral blood after maintenance therapy completion.
Time Frame: At the end of Cycle 2 of induction therapy (each cycle is 28 days), following consolidation phase (after 6 cycles of induction, consolidation is 4 weekly doses of obinutuzumab), within 30 days of completing protocol therapy (up to 15 months total)
Population: one participant died during the Induction Phase
Measure: Count of Participants; unit: Participants
Arm/Group | Bendamustine + Obinutuzumab (BO)
Number analyzed (Participants) | 20
Participants
  MRD negative (blood) after Induction Phase | 13
  MRD negative (blood and marrow) post-Consolidation Phase | 10
  MRD negative (blood only) post-Consolidation Phase | 6

3. Secondary Outcome: Estimate the Concordance Rate Between Peripheral Blood (PB) and Bone Marrow Aspirates (BMA) in Predicting MRD Status.
Description: Concordance between PB and BMA in predicting MRD negative status will be summarized by percent of subjects in which MRD status is concordant (i.e., both positive in the PB and BMA or both negative in the PB and BMA).
Time Frame: At the end of Cycle 2 of induction therapy (each cycle is 28 days), following consolidation phase of therapy (after 6 cycles of induction, consolidation is 4 weekly doses of obinutuzumab), and within 30 days of completing protocol therapy
Population: one participant died during the Induction Phase
Measure: Count of Participants; unit: Participants
Arm/Group | Bendamustine + Obinutuzumab (BO)
Number analyzed (Participants) | 20
Participants | 14

4. Secondary Outcome: Determine Objective Response Rates (CR + PR) With Induction Bendamustine and Obinutuzumab (BO) in Previously Untreated MCL Using the Lugano Classification for Response in Lymphoma
Description: Lugano criteria will be used to assess radiographic response by CT and/or positron emission tomography (PET) imaging. Imaging for response assessment will be performed after 4 cycles of induction therapy, after consolidation obinutuzumab, and after cycles 4 and 8 of maintenance obinutuzumab. Bone marrow biopsy will be performed verify complete responses. Assessed as the best response over the course of therapy from any of the following time points: at the end of induction cycle 4 (each cycle is 28 days), after consolidation therapy (post-induction, consolidation is 4 weekly doses Obinutuzumab), and after Cycles 4 and 8 of Maintenance Obinutuzumab (each cycle is 8 weeks).
Time Frame: Assessed up to cycle 8 of maintenance therapy, up to 15 months on study
Population: one participant died during the Induction Phase
Measure: Count of Participants; unit: Participants
Arm/Group | Bendamustine + Obinutuzumab (BO)
Number analyzed (Participants) | 20
Participants
  Complete Response | 15
  Partial Response | 4
  Overall Objective Response | 19

5. Secondary Outcome: Overall Survival (OS)
Description: For a given participant, OS will be measured from C1D1 of the induction chemoimmunotherapy to the day the subject dies. Survival times of subjects who are still alive at the end of the follow-up period will be censored. OS will be summarized using point estimate of the median OS, along with the 95% confidence interval.
Time Frame: Up to 3 years
Measure: Number (95% Confidence Interval); unit: percent participants
Arm/Group | Bendamustine + Obinutuzumab (BO)
Number analyzed (Participants) | 21
percent participants
  2-year Overall Survival | 75.4 [50.6 to 89.0]
  3-year Overall Survival | 60.9 [33.9 to 79.7]

6. Secondary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v5.0 During Therapy Induction BO Chemoimmunotherapy and Obinutuzumab Consolidation and Maintenance
Description: Count of toxicities from the initiation of study treatment until 30 days following the last administration of study treatment or study discontinuation/termination; after this period, only serious adverse events (SAEs) that are possibly, probably, or definitely attributed will be reported. For a given subject, toxicities will be assessed from the time of C1D1 of study therapy until 30 days after completion of final dose of study-related treatment.
Time Frame: Up to 25 months (until 30 days after completion of final dose of study-related treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Bendamustine + Obinutuzumab (BO)
Number analyzed (Participants) | 21
Participants | 21

7. Post Hoc Outcome: Progression Free Survival (PFS) at 3 Years
Description: For each patient, progression-free survival (PFS) will be measured from C1D1 of induction chemoimmunotherapy to the day patient experiences an event of disease progression or death, whichever occurs first. If a patient has not experienced an event at the time of analysis, patient's data will be censored at the date of the last available evaluation. The 3-year PFS probability will be estimated using the Kaplan-Meier method. From the date of C1D1 of induction therapy to the date of progression or death; in the absence of progression or death, subjects will be followed for a minimum of 24 months after completion of study-related treatment. PFS rates at 3 years are reported here.
Time Frame: Up to 3 years
Measure: Number (95% Confidence Interval); unit: percent participants
Arm/Group | Bendamustine + Obinutuzumab (BO)
Number analyzed (Participants) | 21
percent participants | 58.7 [33.2 to 77.3]

ADVERSE EVENTS:
Time Frame: up to 36 months
Arm/Group | Bendamustine + Obinutuzumab (BO)
All-Cause Mortality (participants affected / at risk) | 9/21
Serious Adverse Events (participants affected / at risk) | 9/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bendamustine + Obinutuzumab (BO) (N=21)
Atrial fibrillation / flutter (Blood and lymphatic system disorders) | 2 (2)
Myocardial infarction (Cardiac disorders) | 1 (1)
Colitis / Abdominal Infection (Gastrointestinal disorders) | 2 (2)
Infusion related reaction (General disorders) | 2 (2)
Allergic reaction (Immune system disorders) | 1 (1) — possible drug reaction - Bactrim
Pneumonia (Infections and infestations) | 2 (3)
Thrombocytopenia (Investigations) | 1 (1)
Neutropenia (Investigations) | 1 (2) — occurred outside of the time frame of when neutropenia would be an expected treatment-related toxicity
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (6) — 1 subject colon adenocarcinoma, 1 subject experienced 3 events: melanoma in situ, squamous cell carcinoma, and basal cell carcinoma, 1 subject squamous cell carcinoma, 1 subject with increasing size of retrobulbar (brain) mass
Genital Edema (Reproductive system and breast disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bendamustine + Obinutuzumab (BO) (N=21)
Anemia (Blood and lymphatic system disorders) | 4 (10)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (2)
Palpitations (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (2)
Hypothyroidism (Endocrine disorders) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 2 (2)
Dry eye (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 7 (11)
Diarrhea (Gastrointestinal disorders) | 10 (15)
Dry mouth (Gastrointestinal disorders) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 4 (6)
Dysphagia (Gastrointestinal disorders) | 1 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (4)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 12 (23)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (8)
Chills (General disorders) | 1 (1)
Edema limbs (General disorders) | 3 (4)
Fatigue (General disorders) | 11 (24)
Fever (General disorders) | 4 (5)
Flu like symptoms (General disorders) | 2 (2)
General disorders and administration site conditions - Other, specify (General disorders) | 7 (15)
Localized edema (General disorders) | 2 (3)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 4 (6)
Cytokine release syndrome (Immune system disorders) | 2 (4)
Fever (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (3)
Soft tissue infection (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3)
Vaginal infection (Infections and infestations) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (2)
Bruising (Injury, poisoning and procedural complications) | 3 (3)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (4)
Blood lactate dehydrogenase increased (Investigations) | 1 (7)
Creatinine increased (Investigations) | 1 (3)
Investigations - Other, specify (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 9 (35)
Neutrophil count decreased (Investigations) | 10 (28)
Platelet count decreased (Investigations) | 6 (8)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 2 (4)
White blood cell decreased (Investigations) | 10 (33)
Anorexia (Metabolism and nutrition disorders) | 4 (5)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (9)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (3)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (10)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4)
Dizziness (Nervous system disorders) | 2 (4)
Dysgeusia (Nervous system disorders) | 5 (5)
Headache (Nervous system disorders) | 2 (2)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (3)
Syncope (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (2)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (7)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (11)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 (3)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 5 (11)
Hypotension (Vascular disorders) | 3 (3)
Phlebitis (Vascular disorders) | 2 (2)
Thromboembolic event (Vascular disorders) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-13): https://cdn.clinicaltrials.gov/large-docs/26/NCT03311126/Prot_SAP_000.pdf